CLINICAL TRIAL: NCT06121505
Title: Low-dose Radiation Therapy and Stereotactic Body Radiation Therapy Combined With PD-1 Inhibitor Sintilimab and Chemotherapy Versus PD-1 Inhibitor Combined With Chemotherapy as First-line Treatment for Patients With Locally Advanced or Metastatic Squamous Cell Lung Cancer: A Randomized, Phase II Multicenter Clinical Trial
Brief Title: Phase II Trial: Low-Dose Radiation + SBRT + Sintilimab + Chemotherapy vs. Sintilimab + Chemotherapy in Locally Advanced or Metastatic Squamous Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Division of Thoracic Tumor Multimodality Treatment, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHC-002
Record Dates: First submitted 2023-10-31; First posted 2023-11-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Squamous Cell Carcinoma
Keywords: SBRT; Immunotherapy; LDRT; Lung Squamous Cell Carcinoma
MeSH Terms: interventions — Radiotherapy; Radiosurgery; Drug Therapy; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy combined with sintilimab and chemotherapy (Experimental): Subjects received radiotherapy (SBRT+LDRT). Sintilimab combined with standard platinum-containing double-drug chemotherapy was performed within 1 week after the end of radiotherapy.
  Interventions: Radiation: low-dose radiation therapy and stereotactic body radiation therapy; Drug: chemotherapy; Drug: Sintilimab
- Sintilimab+Chemotherapy (Active Comparator): Subjects received sintilimab combined with standard platinum-based doublet chemotherapy for a total of 4 cycles.
  Interventions: Drug: chemotherapy; Drug: Sintilimab

INTERVENTIONS:
Radiation: low-dose radiation therapy and stereotactic body radiation therapy — Patients will receive radiation therapy.
  Other Names: RT
  Arms: Radiotherapy combined with sintilimab and chemotherapy
Drug: chemotherapy — Patients will receive sintilimab combined with standard platinum-based doublet chemotherapy for a total of 4 cycles. Patients subsequently received maintenance treatment with sintilimab, and continued treatment until disease progression (PD), intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor treatments, death, or other circumstances that should stop treatment as specified in the protocol. Whichever occurs first. The maximum treatment time with sintilimab is 24 months (or 35 cycles).
  Other Names: standard platinum-containing double-drug chemotherapy
Drug: Sintilimab — Patients will receive sintilimab combined with standard platinum-based doublet chemotherapy for a total of 4 cycles. Patients subsequently received maintenance treatment with sintilimab, and continued treatment until disease progression (PD), intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor treatments, death, or other circumstances that should stop treatment as specified in the protocol. Whichever occurs first. The maximum treatment time with sintilimab is 24 months (or 35 cycles).

SUMMARY:
This is a randomized, controlled, open-label, multicenter phase II clinical trial comparing the efficacy and safety of low-dose radiation therapy and stereotactic body radiation therapy combined with PD-1 inhibitor (sintilimab) and standard platinum-based doublet chemotherapy versus PD-1 inhibitor (sintilimab) combined with standard platinum-based doublet chemotherapy as first-line treatment in patients with locally advanced or metastatic squamous cell lung cancer.

There will be 57 subjects in the experimental group and 57 subjects in the control group, with a total of 114 subjects.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter phase II clinical trial comparing the efficacy and safety of low-dose radiation therapy and stereotactic body radiation therapy combined with PD-1 inhibitor (sintilimab) and standard platinum-based doublet chemotherapy versus PD-1 inhibitor (sintilimab) combined with standard platinum-based doublet chemotherapy as first-line treatment in patients with locally advanced or metastatic squamous cell lung cancer. Patients with previously untreated, locally advanced or metastatic (unresectable or not eligible for definitive chemoradiotherapy, stage IIIB-IV) squamous cell lung cancer who have signed informed consent will be screened for eligibility. Qualified subjects who meet the inclusion criteria will be randomly assigned at a 1:1 ratio to the experimental group (radiation therapy plus sintilimab and chemotherapy) or the control group (sintilimab plus chemotherapy). Based on sample size estimation according to statistical hypotheses, there will be 57 subjects in the experimental group and 57 subjects in the control group, with a total of 114 subjects. Subjects in the experimental group will receive radiation therapy. Within 1 week after radiation therapy, they will receive treatment with sintilimab combined with standard platinum-based doublet chemotherapy. Chemotherapy combined with immunotherapy will consist of a total of 4 cycles. Patients will subsequently receive maintenance therapy with sintilimab. Subjects in the control group will receive treatment with sintilimab combined with standard platinum-based doublet chemotherapy, consisting of a total of 4 cycles. Patients will subsequently receive maintenance therapy with sintilimab. The primary efficacy endpoint of this study is objective response rate (ORR), as assessed by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 75 years old;
2. Histologically or cytologically confirmed squamous cell lung cancer, imaging confirmed locally advanced or metastatic disease (unresectable or not eligible for definitive chemoradiotherapy, stage IIIB-IV);
3. According to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), there is at least one imaging measurable lesion;
4. Enough to provide quality control qualified tumor tissue or cell wax blocks to detect PD-L1 expression;
5. Have not received any systemic anti-tumor treatment for locally advanced or metastatic disease in the past;

Exclusion Criteria:

1. The pathology is small cell lung cancer (SCLC), including lung cancer mixed with SCLC and non-small cell lung cancer (NSCLC)；
2. The pathology is lung adenocarcinoma, including lung cancer mixed with lung adenocarcinoma and lung squamous cell carcinoma;
3. EGFR gene sensitive mutation or ALK fusion positive or ROS1 fusion positive;
4. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or another drug that stimulates or synergistically inhibits T cell receptors;
5. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Every 6 weeks (±7 days) from the first dose of study drug, and every 12 weeks (±7 days) after 48 weeks (up to 24 months).
  The proportion of subjects with complete response (CR) or partial response (PR) in the analyzed population as judged by the investigator according to RECIST v1.1 criteria. ORR = (number of subjects with CR + PR) / total number of subjects * 100%.

SECONDARY OUTCOMES:
6-month PFS rate | From date of randomization to 6 months.
  The 6-month PFS rate is defined as the proportion of patients who did not experience disease progression or death from any cause at the time of 6 months.
1-year PFS rate | From date of randomization to 1 years.
  The 1-year PFS rate is defined as the proportion of patients who did not experience disease progression or death from any cause at the time of 1 year.
overall survival(OS) | From date of randomization to the time when the subject died from any cause, assessed up to 36 months.
  OS is defined as the time from randomization to the death of the subject from any cause.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Progression-free survival (PFS) is defined as the time from randomization to first imaging disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (6):
- China (6):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hunan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang R, Chen M, Yin N, Xue J. Low-dose radiation and stereotactic body radiotherapy with PD-1 inhibitor sintilimab and chemotherapy for first-line treatment of locally advanced or metastatic squamous lung cancer: protocol for a randomised phase II trial (IHC002 study). BMJ Open. 2025 Aug 31;15(8):e094859. doi: 10.1136/bmjopen-2024-094859. PMID 40887121